CLINICAL TRIAL: NCT06621394
Title: The Effect of Mediterranean Diet and Mindfulness Eating on Depression Severity in People With Obesity and Major Depressive Disorder - a Randomized Controlled Study With Mulitfactorial Design
Brief Title: The Effect of Mediterranean Diet and Mindfulness Eating on Depression Severity in People With Obesity and Major Depressive Disorder
Acronym: MEDIMIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Robert Bosch Center for Integrative Medicine and Health (Unknown); Department of Psychosomatic Medicine, Robert Bosch Hospital Stuttgart (Unknown); Microbial Genetics, Interfaculty Institute of Microbiology and Infection Medicine Tübingen, University of Tübingen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: medimind
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-11

CONDITIONS: Depressive Disorder, Major
Keywords: depression; mediterranean diet; mindfulnes eating; nutrition; obesity
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Obesity

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Who Masked: Outcomes Assessor
Masking Description: data analysis will be conducted blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mediterranean Diet (Experimental)
  Interventions: Other: nutritional intervention
- Mindful Eating (Experimental)
  Interventions: Behavioral: Mindful Eating
- Mediterranean Diet and Mindful Eating (Experimental)
  Interventions: Other: nutritional intervention; Behavioral: Mindful Eating
- Befriending (Sham Comparator)
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: nutritional intervention — nutritional intervention to mediterranean diet
  Arms: Mediterranean Diet; Mediterranean Diet and Mindful Eating
Behavioral: Mindful Eating — intervention regarding mindful eating, e.g. attention while eating, apprechiation of food
  Arms: Mediterranean Diet and Mindful Eating; Mindful Eating
Other: Attention Control — Befreinding Control Group: Provision of same amout of time and attention, without having an intervention, e.g. talking about hobbies and interests, playing card games
  Arms: Befriending

SUMMARY:
The present study investigates the effect of Mediterranean Diet and Mindful Eating on depression severity in people with obesity and major depressive disorder. The factorial design allows to investigate potential synergistic effects of the interventions. Participants will be randomized to one of the four intervention groups (mediterranean diet, mindful eating, their combination and a befriending control group). The intervention consists of a 12-week period, followed by a 12-week follow up. The primary outcome is depression severity.

DETAILED DESCRIPTION:
Depression and obesity are highly prevalent diseases that are strongly correlated. There is a growing gap in care and treatment options for those affected. The effectiveness of a Mediterranean Diet on mental health has already been shown in various studies. Additionally to physiological effects of nutrient intake, also the psychological factor of changing the way of eating seem to play a role. The present study investigates the effect of a Mediterranean Diet and Mindful Eating on depression severity in people with obesity and clinically diagnosed major depressive disorder. The factorial design allows to investigate potential synergistic effects of the interventions. Participants will be randomized to one of the four intervention groups (mediterranean diet, mindful eating, their combination and a befriending control group). The intervention consists of a 12-week period, where five individual nutrition consueling meetings will take place, followed by a 12-week follow up. The primary outcome is depression severity. Secondary outcomes and analyzes include quality of life, self-efficacy, mediterranean diet and mindfulness eating scores, anthropometric measurements, as well as mediator and moderator analysis, a microbiome analysis, a qualitative evaluation and an economic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of clinically diagnosed major depression
* At least moderate depression severity: BDI-II ≥ 20
* obesity: BMI ≥ 30 kg/m2
* Stable co-intervention: no change in the type, dosage or frequency of antidepressant medication and/or psychotherapy four weeks before and during the study
* Low adherence to the mediterranean diet: MEDAS < 10
* Low adherence to mindful eating: MEI < 5.13

Exclusion Criteria:

* Diseases of the gastrointestinal tract that do not allow adequate implementation of the intervention (e.g. irritable bowel syndrome, post-bariatric surgery, colorectal carcinoma)
* Metabolic diseases with strong impact on intervention (e.g. type 1 diabetes mellitus, chronic kidney disease)
* Severe food allergies and intolerances, that do not allow adequate implementation of the intervention
* Diagnosed, current psychological comorbidities (bipolar disorder, eating disorder, personality disorder, psychosis)
* intake of antibiotics in the last three months current substance abuse
* Pregnancy and breatfeeding
* Suicidal ideation
* unable to participate or complete questionnaires

Healthy Volunteers:

samples of 32 healthy volunteers are included for microbiome analysis only (

inclusion criteria:

* age ≥ 18 years
* BMI 20 - 30 kg/m^2

exclusion criteria:

* depression or other psychological comorbidities (bipolar disorder, eating disorder, personality disorder, psychosis)
* high adhernece to mediterranean diet: MEDAS ≥ 10
* high adherence to mindful eating: MEI ≥ 5.13
* Diseases of the gastrointestinal tract or metabilic diseases (e.g. irritable bowel syndrome, post-bariatric surgery, colorectal carcinoma, type 1 diabetes mellitus)

  -- intake of antibiotics in the last three months current substance abuse
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Depression severity | 12 weeks
  Beck Depression Inventory - II (BDI-II) scores range from 0 to 63 with higher scores indicating higher depression severity

SECONDARY OUTCOMES:
Depression severity, self assessment | 24 weeks
  Beck Depression Inventory - II (BDI-II) scores range from 0 to 63 with higher scores indicating higher depression severity
Depression Remission Rates | 12 weeks, 24 weeks
  rates of participants showing no depressive symptoms, defined as BDI-II less than 9
Quality of Life | 12 weeks, 24 weeks
  Short Form-36 Health Survey (SF-36), mental and physical sum score, which can be further divided into the subscales vitality, physical functioning, physical pain, general health perception, physical role function, emotional role function, social role function and psychological well-being, higher scores indicate a higher quality of life
Self-efficacy | 12 weeks, 24 weeks
  general self-efficacy expectation scale, score ranges from 10 to 40, with a higher score indicating a greater expectation of self-efficacy
Health status | 12 weeks,
  European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L), results in a 5-digit number that describes the patient's health state
Adhernece to Mediterranean Diet | 12 weeks, 24 weeks
  mediterranean diet adherence score (MEDAS) scores range from 0 to 14 with higher values indicating higher adherence to mediterranean diet
Adherence to Mindfulnes Eating | 12 weeks, 24 weeks
  Mindfulness Eating Inventory (MEI), score ranges from 1 to 6, with higher scores indicating higher adherence to mindfulness eating
Depression severity, rater assesment | 12 weeks
  Depresion severity is assessed by psychologists by using the MARDS tool. Scores range from 0 to 60 with higher scores idnicating higher severity of depression
BMI | 12 weeks, 24 weeks
  weight and height will be combined to report BMI in kg/m^2
Waist to Hip ratio | 12 weeks, 24 weeks
  ratio of weight circumference and hip circumference
Body composition: muscle mass | 12 weeks, 24 weeks
  muscle mass as a percentage of body weight
Body composition: fat mass | 12 weeks, 24 weeks
  fat mass as a percentage of body weight
adverse events | 12 weeks, 24 weeks
  time point, duration (in hours or days) and strengths (on a scale from one to ten) of andverse events will be assessed as well as perception of connection between occurrence of adverse event and the intervention
Microbiome Analysis | 12 weeks
  16s RNA sequencing
cost-utility analysis | 12 weeks
  from EQ-5D-5L values quality adjustes life years (QUALYS) will be calulated to conduct cost-utility analysis from participants perspective
Qualitative evaluation | 12 weeks
  Semi-structured interviews will consider two areas:
  1. the perception on the intervention in terms of feasibility, difficulties in implementation, perception of study setting, planning of long-term implementation, etc.
  2. perception of effects of interventions, qualitative evaluation of changes in outcoms, i.e. mood, psychological and physical well-being, self-efficacy, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Bosch Center for Integrative Medicine and Health, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No